CLINICAL TRIAL: NCT04173026
Title: Dissemination and Implementation of Stroke Prevention Looking at the Care Environment (DISPLACE) Part 3
Brief Title: Dissemination and Implementation of Stroke Prevention Looking at the Care Environment
Acronym: DISPLACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Julie Kanter, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NIH 5R01HL133896-02
Record Dates: First submitted 2019-11-15; First posted 2019-11-21 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Randomized cluster controlled implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider intervention (Active Comparator): A web-based application called ProviderMinder has been developed and will be used to alert providers when a patient who has been lost-to-follow-up or has missed their Sickle Stroke Screen (TCD). This will allow providers to follow up with such patients and improve screening rates.
  Interventions: Other: Provider-level intervention
- Provider and Patient level intervention (Active Comparator): A web-based application called ProviderMinder has been developed and will be used to alert providers when a patient who has been lost-to-follow-up or has missed their Sickle Stroke Screen (TCD). This will allow providers to follow up with such patients and improve screening rates. Additionally, sites will have a patient intervention of a single Sickle Stroke Screen coordinator who will interact directly with patients to schedule, reschedule, remind, and follow-up on stroke screening. This person will also act as a point of contact for any educational needs the patient may have. The second patient intervention will include the caregivers own mobile device. When Sickle Stroke Screens are scheduled the coordinator will ensure these appointments are directly put into the caregiver's mobile device calendar acting as an additional reminder for stroke screening.
  Interventions: Other: Provider-level intervention; Other: Patient-level intervention

INTERVENTIONS:
Other: Provider-level intervention — Provider minder is a provider-based scheduling and reminder system for stroke screening in SCD
  Other Names: Provider Minder
Other: Patient-level intervention — 50% of centers are randomized to a single stroke screen coordinator as the point of contact for sickle stroke screen
  Other Names: Single Coordinator
  Arms: Provider and Patient level intervention

SUMMARY:
The Dissemination and Implementation of Stroke Prevention Looking at the Care Environment (DISPLACE) study is a multi-center, national, National Heart, Lung and Blood Institute (NHLBI)-funded grant to look at the real-world implementation of stroke prevention guidelines (STOP Protocol) in which transcranial Doppler (TCD), a measure of cerebral blood vessel velocity, is used to screen for stroke risk in children ages 2-16 with sickle cell anemia (SCA). Part 3 of the DISPLACE study is an implementation clinical trial designed to test novel implementation strategies with the goal of improving adherence and implementation of stroke screening. 16 of the lowest scoring implementation rates from DISPLACE Part 1 will participate in DISPLACE Part 3. All original 28 sites from DISPLACE Parts 1 and 2 will receive a patient and provider educational intervention including a re-branding of the TCD as "Sickle Stroke Screen" with a new infographic and educational materials. The 16 sites with moving to Part 3 will be provided a Provider reminder strategy, which is a web based application designed to remind providers of when patients are due for their Sickle Stroke Screen. These 16 sites will be randomized and 8 will be given an additional Patient Communication Strategy. These sites will have a single designed coordinator with whom patients will communicate with about scheduling, rescheduling, and any other questions regarding their Sickle Stroke Screen. Upon completion, data will be analyzed to compare those who have had TCD screenings done appropriately and those who did not as well as the overall effect of the multi level interventions on the changes in TCD rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell anemia (SCA) identified at each institution through International Classification of Diseases 9/10 (ICD-9/ICD-10) codes and local patient databases.
* Patients must have been seen by the designated institution (documented in medical record) a minimum of two times in the either inpatient or outpatient setting at the institution between the years of 01/01/2018-12/31/2019.
* Patients identified will include those currently aged 2-7. Thus children born from 2012 and onward.
* Patients already receiving primary or secondary stroke prevention therapy with CRCT will be included in registration in Web Data Coordination Unit (WEBDCU) but not included in PROVIDER MINDER as they do not require ongoing TCD/SICKLE STROKE SCREEN based on protocol.

Exclusion Criteria:

* Patients who do not have SCA
* Patients who were born before 2012 and therefore do not meet age criteria.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
1. Change in uptake and use of the stroke prevention guidelines (STOP Protocol) as defined in the NHLBI (National Heart, Lung, and Blood Institute) 2014 Sickle Cell Disease (SCD) Guidelines by assessing stroke risk with yearly TCD screens | baseline-2 years
  The TCD measures the speed of blood flow in the blood vessels of the brain. Any unusually slow of fast speed may indicate a child is at a higher risk for stroke. By ensuring patients receive a yearly TCD more children will get a proper intervention and ideally prevent stroke.
2. Change in uptake and use of the stroke prevention guidelines (STOP Protocol) as defined in the NHLBI 2014 SCD Guidelines by implementing chronic red cell transfusion (CRCT) in patients noted to have abnormal TCD screens. | baseline-2 years
  CRCT has been shown to severely decrease the incidence of stroke in patients who have had TCD screenings with an abnormal result.
Change in uptake and use of the stroke prevention guidelines (STOP Protocol) as defined in the NHLBI (National Heart, Lung, and Blood Institute) 2014 SCD (Sickle Cell Disease) Guidelines by re-screening patients with conditional TCD screens | baseline-2 years
  Patients who have a condition TCD are considered to of slightly higher risk than patients with a normal TCD. By re-screening these patients in a shorter time period, providers are able to confirm or reject the initial screening and make the best plan for stroke prevention depending on these outcomes.
A difference in uptake and use of the stroke prevention guidelines (STOP Protocol) as defined in the NHLBI 2014 SCD Guidelines between between implementation arms measured by assessing yearly TCD screening rates. | baseline-2 years
  Any difference in TCD implementation rates between each intervention arms will help determine optimal implementation procedures.

SECONDARY OUTCOMES:
Barriers to obtaining TCD screening | baseline-2 years
  Participating sites will carry out key informant interviews with patients/caregivers and stakeholders will be analyzed using content analysis to identify themes pertaining to barriers to obtaining TCD screening, as well as overall perceptions of the intervention(s), barriers to implementing the intervention(s) and satisfaction with the intervention(s).
Enablers to obtaining TCD screening | baseline - 2 years
  Participating sites will carry out key informant interviews with patients/caregivers and stakeholders will be analyzed using content analysis to identify themes pertaining to enablers to obtaining TCD screening, as well as overall perceptions of the intervention(s), enablers to implementing the intervention(s) and satisfaction with the intervention(s).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kanter, MD, Principal Investigator — University of Alabama at Birmingham
Locations (15):
- United States (15):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Nemours Center for Cancer & Blood Disorders, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Shands Children's Hospital, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Children's Heathcare of Atlanta, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Vidant Medical Center, Greenville, North Carolina
  - Vanderbilt Children's Hospital, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
To be determined.

REFERENCES:
- [Derived] Schlenz AM, Phillips SM, Mueller M, Humphrey D, Stevens J, Williams LP, Nickel RS, Dolatshahi L, Miller RE, Hulbert ML, Lee MT, Alvarez O, Fuh B, McNaull MA, Bhasin N, Melvin CL, Adams RJ, Kanter J. Successful implementation of stroke risk screening for sickle cell anemia in the DISPLACE study: results of a cluster randomized trial. Implement Sci. 2025 Nov 26;20(1):50. doi: 10.1186/s13012-025-01462-3. PMID 41299691